CLINICAL TRIAL: NCT03822884
Title: Pharmacokinetic/Pharmacodynamic Study of 3 Subcutaneous Single Dose Epoetin Alfa Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio Sidus SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HMX.1.003
Record Dates: First submitted 2016-11-11; First posted 2019-01-30 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hemax® PFS 40,000 UI (Experimental): Epoetin Alfa 40000 UNT/ML subcutaneous single dose
  Interventions: Drug: Epoetin Alfa 40000 UNT/ML
- Hemax® 40,000 UI (Experimental): Epoetin Alfa 40000 UNT/ML subcutaneous single dose
  Interventions: Drug: Epoetin Alfa 40000 UNT/ML
- Erypo ® 40,000 UI (Active Comparator): Epoetin Alfa 40000 UNT/ML subcutaneous single dose
  Interventions: Drug: Epoetin Alfa 40000 UNT/ML

INTERVENTIONS:
Drug: Epoetin Alfa 40000 UNT/ML — 40.000 UI subcutaneous single dose
  Other Names: Hemax; Hemax PFS; Erypo

SUMMARY:
Pharmacokinetic/Pharmacodynamic Study of 3 Epoetin Alfa Formulations in Single Subcutaneous Doses Administered to Healthy Volunteers

SPONSOR Biosidus S.A.

DETAILED DESCRIPTION:
TITLE

Pharmacokinetic/ Pharmacodynamic Study of 3 Epoetin Alfa Formulations in Single Subcutaneous Doses Administered to Healthy Volunteers

SPONSOR

Biosidus S.A.

PRINCIPAL INVESTIGATOR

Guillermo Di Girolamo, M.D., National License No. 56857, domiciled at Congreso 3137 (Calle 75), San Andrés (1651), Telephone/Fax: 4753 - 8211, e - mail: gdigirolamo@arnet.com.ar

CO-INVESTIGATORS

Guillermo Alberto Keller, M.D., National License No.106.860, domiciled at Murgiondo 376, CABA. Cell Phone: 1563615376 - e-mail: drguillermokeller@yahoo.com.ar

Paola Czerniuk, M.D., National License No. 84280, domiciled at Paraguay 3559, Piso 6, Dto A, CABA. Cell Phone 1550189563, e - mail: pczerniuk@intramed.net.ar SITE Centro de Medicina Integral S.R.L. - Address: Avenida Belgrano 1844, CABA (C1094) - Telephone: (011) 4383 - 5145

LABORATORY

Laboratorio de Calidad de Biosidus SA - Constitución 4234 (C1254ABX) Buenos Aires, Argentina - Tel. 4909 8000 - Fax 4909 8055

OBJECTIVES

Primary: To compare the pharmacokinetic and pharmacodynamic behavior of three formulations of epoetin alfa after subcutaneous administration of 40,000 UI:

* Erypo ® 40,000 UI, liquid without albumin, prefilled syringe, produced by Janssen - Cilag GmbH (Reference Formulation, "R")
* Hemax® 40,000 UI, lyophilized with albumin, vial, produced by Biosidus SA (Test Formulation Number 1, "T1")
* Hemax® PFS 40,000 UI, liquid without albumin, prefilled syringe, produced by Biosidus SA (Test Formulation Number 2, "T2")

Secondary: To assess the pharmacological action, through quantification of blood reticulocytes at different time points as a surrogate pharmacodynamic marker. Assessment of adverse effects and tolerance.

TRIAL DESIGN

Open, randomized, 3 - arm, cross - over, sequential, and balanced

DISCONTINUATION SCHEME

The sponsor and the investigators can independently discontinue the study at any time if there is a mere possibility of or in case of occurrence of a serious adverse effect or situation that might affect the volunteer's health. If the Hb exceeds 18 g/ dl confirmed by repetition of the analysis at the pre - dose control in each phase, the volunteer will be excluded and 1 unit of blood will be collected. If, after the procedure, it is still above 18 g/ dl, another 0.5 or 1 Unit of blood will be collected, based on medical judgment.

NUMBER OF VOLUNTEERS

24 (twenty - four) at first. Since it is a sequential design, if the statistical analysis of the first 24 volunteers does not show biosimilarity, 12 additional volunteers will be included up to a total of 36 (thirty - six) volunteers.

DURATION OF THE STUDY

3 months

Selection and recruitment period: 2 (two) months

TIME THE STUDY WILL TAKE

Visit I: Selecting volunteers, obtaining informed consents, performing baseline tests.

Visits II, III, and IV: They will consist of 3 hospitalization phases -one for subcutaneous administration of Test Formulation Number 1 (T1), another for subcutaneous administration of Test Formulation Number 2 (T2), and a third one for subcutaneous administration of Reference Formulation (R), with a washout period of no fewer than 28 days between phases.

Sampling times for erythropoietin quantification in each phase, carried out by Biosidus SA, will be: pre - dose and 1, 2, 4, 6, 7, 8, 9, 10, 11, 12, 15, 24, 48, 72, 96, and 120 hours post - dose.

Telephone contact: The Principal Investigator or the healthcare staff assigned by the Principal Investigator will contact the volunteer by phone after the volunteer's discharge until the last (120 - hour) outpatient collection in order to ask about tolerance to the medication and presence of adverse effects.

Blood samples will be collected for red blood cell, Hb, and reticulocyte counting using flow cytometry performed by Biosidus SA, as an erythropoietin surrogate pharmacodynamic marker at the following time points: pre - dose (0 hours), 24, 48, 72, 96, 120, and 240 hours.

Another blood sample will be collected for red blood cell and Hb count after 504 hours (21 days after the dose), 7 days before starting the next treatment cycle, in order to determine whether the volunteer complies with one of the inclusion criteria for the next phase, i.e. not exceeding 18 g/ dl of Hg.

DOSE / ROUTE / REGIME / OF THE INVESTIGATION PRODUCTS

Single 40,000 UI dose of epoetin alfa. The following formulations will be assessed after administering 1 subcutaneous injection on the arm:

* Erypo ® 40,000 UI, liquid without albumin, prefilled syringe, produced by Janssen - Cilag GmbH (Reference Formulation, "R")
* Hemax® 40,000 UI, lyophilized with albumin, vial, produced by Biosidus SA (Test Formulation Number 1, "T1")
* Hemax® PFS 40,000 UI, liquid without albumin, prefilled syringe, produced by Biosidus SA (Test Formulation Number 2, "T2")

There will be 6 randomly assigned sequences:

1. R - T1 - T2
2. R - T2 - T1
3. T1 - R - T2
4. T1 - T2 - R
5. T2 - R - T1
6. T2 - T1 - R

COMPARISON DRUG

Erypo ® 40,000 UI, liquid without albumin, prefilled syringe, produced by Janssen - Cilag GmbH (Reference Formulation, "R")

COMPARATIVE PHARMACOKINETIC AND PHARMACODYNAMIC ASSESSMENT BETWEEN THE FORMULATIONS

Based on the erythropoietin serum concentration results, at the different sampling times, the following variables will be calculated:

* AUC0 - 120h: Area under the serum concentration - time curve 0 - 120 h.
* AUC0 - ∞: Area under the serum concentration - time curve from time 0 extrapolated to infinity (∞).
* Cmax: Maximum serum concentration of erythropoietin.
* Cmin: Minimum serum concentration of erythropoietin.
* Tmax: Time to maximum serum concentration of erythropoietin.

The difference between Tmax times in each test formulations and the reference formulation will be assessed, and the elimination rate constant and half - life of the drug in the body will be calculated.

The average results for each formulation will be presented, as well as each volunteer's individual results.

STATISTICAL ANALYSIS

CALCULATION OF THE SAMPLE SIZE:

The size of the sample (n:24) was established based on literature data and information from absolute and relative bioavailability studies performed with the drug before by Biosidus SA. Since it is a sequential design, if the statistical analysis of the first 24 volunteers does not show biosimilarity, 12 additional volunteers will be included up to a total of 36 (thirty - six) volunteers.

ANALYSIS PLAN

COMPARATIVE PHARMACOKINETIC ANALYSIS BETWEEN FORMULATIONS

* AUCT / AUCR: Quotient between the area under the curve of the TEST formulation and the area under the curve of the REFERENCE. For the log transformation, the 90% confidence interval of the AUC ratio (for AUC0 - 120h and AUC0 - ∞) should be within the range of 0.80 - 1.25.
* CmaxT / CmaxR: Quotient between the Cmax of the Test formulation and the Cmax of the Reference. For the log transformation, the 90% confidence interval of the Cmax ratio should be within the range of 0.80 - 1.25.

COMPARATIVE PHARMACODYNAMIC ANALYSIS BETWEEN THE FORMULATIONS

* Maximum number of reticulocytesT / Maximum number of reticulocytesR: Quotient between the maximum number of reticulocytes in the Test formulation and the maximum number of reticulocytes in the Reference.

Using ANOVA, the possible differences between subjects, treatments, and periods will be analyzed.

Outliers: In order to determine possible outliers, a selective - statistical method will be applied.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subjects of both sexes aged 21 - 55 years old.
2. Baseline Hb levels between 11 and 14 in women and between 12 and 15 g/ dl in men.
3. Body Mass Index (BMI) between 19 and 27 kg/ m2.
4. Volunteers whose additional tests (ECG, blood, and urine), performed before their inclusion, are within the normal limits and/ or with no clinical significance based on the investigator's judgment. Women of childbearing potential should have a negative pregnancy test and use a safe contraceptive method during the study (UID or a similarly effective method).
5. Subjects with systolic blood pressure higher than 100 mm Hg and lower than 139 mm Hg, diastolic blood pressure higher than 70 mm Hg and lower than 89 mm H, heart rate higher than 50 and lower than 90 heartbeats per minute after 5 minutes in sitting position and then in standing position (extreme values included).
6. Volunteers who are well disposed to the study and have signed the approved informed consent before the beginning of the study.

EXCLUSION CRITERIA:

1. History of clinically significant allergies (except untreated asymptomatic seasonal allergies).
2. Decrease of more than 20 mm Hg in systolic blood pressure or more than 10 mm Hg in diastolic blood pressure within the first 3 minutes after the change in body position.
3. Volunteers who are or have been taking other drugs (prescription or over - the - counter) within two weeks before the study.
4. Volunteers with a history of autoimmune diseases.
5. Organic CNS, psychological, or psychiatric disorders: epilepsy, manic - depressive tendencies, serious depressive episodes, insomnia, changes in personality.
6. Active infections.
7. Having received live or killed virus or bacteria vaccines within a month before inclusion.
8. Allergic to epoetin alfa or related substances, to human albumin, or any of the ingredients of the formulations.
9. Previous exposure to recombinant epoetin.
10. Active smoker (more than 10 cigarettes/ day).
11. Current clinical evidence of severe digestive disorders.
12. Current clinical evidence of kidney diseases.
13. Current evidence of liver disorders.
14. Current clinical evidence of respiratory or heart diseases.
15. Diabetes mellitus, thyroid dysfunction, or other endocrine disorders.
16. Evidence of active gastroduodenal disease.
17. History of peripheral thrombotic events.
18. An underlying neurological disorder.
19. Current presence of a malignant disease.
20. History of drug or alcohol abuse or addiction within the past three years.
21. History of drug or alcohol abuse within the past two years.
22. Participation in a clinical study within the past three months.
23. A subject who donated or lost blood within three months before the beginning of the study, or who intends to donate blood within three months after the end of the study.
24. Heavy drinker of tea, cocoa, mate, coffee, and/ or caffeinated drinks (> 5 cups/ day) or alcohol (> 50 ml/ day).
25. Electrocardiogram abnormalities.
26. Positive HIV, hepatitis B, or hepatitis C serological testing.
27. Abnormal clinical laboratory results (considered as clinically significant by the physician).
28. Volunteers who have received oral iron supplements within the last month.
29. If Hb exceeds 18 g/ dl on the 504 - hour control before each treatment phase, confirmed by repetition of the analysis.
30. Women who do not use an effective contraceptive method (IUD, condom).
31. Pregnancy and breastfeeding.
32. Uncooperative volunteer.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemax PFS - Hemax - Eprex: Volunteers in this groups received
  1. st Period: 40,000 UI (SC) of Hemax PFS (liquid formulation, without Albumin)
  2. nd Period: 40,000 UI (SC) of Hemax (lyophilized)
  3. rd Period: 40,000 UI (SC) of Eprex/Erypo (reference rhEPO)
- Hemax PFS - Eprex - Hemax: Volunteers in this groups received
  1. st Period: 40,000 UI (SC) of Hemax PFS (liquid formulation, without Albumin)
  2. nd Period: 40,000 UI (SC) of Eprex/Erypo (reference rhEPO)
  3. rd Period: 40,000 UI (SC) of Hemax (lyophilized)
- Hemax - Hemax PFS - Eprex: Volunteers in this groups received
  1. st Period: 40,000 UI (SC) of Hemax (lyophilized)
  2. nd Period: 40,000 UI (SC) of Hemax PFS (liquid formulation, without Albumin)
  3. rd Period: 40,000 UI (SC) of Eprex/Erypo (reference rhEPO)
- Hemax - Eprex - Hemax PFS: Volunteers in this groups received
  1. st Period: 40,000 UI (SC) of Hemax (lyophilized)
  2. nd Period: 40,000 UI (SC) of Eprex/Erypo (reference rhEPO)
  3. rd Period: 40,000 UI (SC) of Hemax PFS (liquid formulation, without Albumin)
- Eprex - Hemax PFS - Hemax: Volunteers in this groups received
  1. st Period: 40,000 UI (SC) of Eprex/Erypo (reference rhEPO)
  2. nd Period: 40,000 UI (SC) of Hemax PFS (liquid formulation, without Albumin)
  3. rd Period: 40,000 UI (SC) of Hemax (lyophilized)
- Eprex - Hemax - Hemax PFS: Volunteers in this groups received
  1. st Period: 40,000 UI (SC) of Eprex/Erypo (reference rhEPO)
  2. nd Period: 40,000 UI (SC) of Hemax (lyophilized)
  3. rd Period: 40,000 UI (SC) of Hemax PFS (liquid formulation, without Albumin)
Period: Overall Study
Arm/Group | Hemax PFS - Hemax - Eprex | Hemax PFS - Eprex - Hemax | Hemax - Hemax PFS - Eprex | Hemax - Eprex - Hemax PFS | Eprex - Hemax PFS - Hemax | Eprex - Hemax - Hemax PFS
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemax PFS - Hemax - Eprex | Hemax PFS - Eprex - Hemax | Hemax - Hemax PFS - Eprex | Hemax - Eprex - Hemax PFS | Eprex - Hemax PFS - Hemax | Eprex - Hemax - Hemax PFS | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.25 (12.71) | 44.25 (0.96) | 41.50 (13.77) | 37.50 (8.96) | 32.25 (12.69) | 41.50 (10.66) | 39.54 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 1 | 2 | 9
  Male | 3 | 2 | 3 | 2 | 3 | 2 | 15
Weight [Mean (Standard Deviation); unit: kg] | 76.00 (14.02) | 72.00 (8.68) | 74.00 (6.32) | 74.25 (8.73) | 69.25 (11.93) | 72.00 (10.20) | 72.92 (9.36)
Height [Mean (Standard Deviation); unit: cm] | 177.50 (15.20) | 127.25 (4.79) | 173.25 (3.95) | 171.00 (13.74) | 171.00 (6.83) | 170.50 (8.54) | 172.58 (9.02)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.01 (2.03) | 24.21 (1.63) | 24.67 (2.21) | 25.44 (1.33) | 23.39 (2.29) | 24.64 (1.33) | 24.39 (1.76)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t
Description: AUC0-t: Area under the serum concentration curve from time 0 to time t (in this case, 120 hours).
Time Frame: 120 h
Measure: Mean (Standard Deviation); unit: mUI*h/mL
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 23 | 24
mUI*h/mL | 37440.71 (16821.67) | 34483.73 (13513.69) | 41150.49 (17095.44)

2. Primary Outcome: AUC0-∞
Description: AUC0-∞: Area under the serum concentration curve resulting from extrapolation from time 0 to time ∞.
Time Frame: 120hr
Measure: Mean (Standard Deviation); unit: mUI*h/mL
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 23 | 24
mUI*h/mL | 42487.04 (19533.78) | 36907.41 (14363.66) | 43978.39 (18786.74)

3. Primary Outcome: Cmax
Description: Cmax: maximum serum concentration of epoetin alfa.
Time Frame: 120hr
Measure: Mean (Standard Deviation); unit: mUI / ml
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 23 | 24
mUI / ml | 853.11 (386.49) | 808.29 (338.10) | 913.07 (429.19)

4. Primary Outcome: Tmax
Description: Tmax: time to the maximum serum concentration of epoetin alfa
Time Frame: 120hr
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 23 | 24
h | 14.17 (5.53) | 15.04 (5.13) | 14.96 (5.16)

5. Secondary Outcome: Reticulocyte Response: Cmax
Description: Reticulocyte count by flow cytometry, as a surrogate marker of the pharmacodynamics of erythropoietin. Maximum reticulocyte concentration achieved.
Time Frame: 120hr
Measure: Mean (Standard Deviation); unit: mUI / ml
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 23 | 24
mUI / ml | 1.23 (0.46) | 1.33 (0.49) | 1.31 (0.48)

6. Secondary Outcome: Reticulocyte Response: AUC 0-120h
Time Frame: 120hr
Measure: Mean (Standard Deviation); unit: mUI*h/mL
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 23 | 24
mUI*h/mL | 341.65 (162.98) | 344.49 (132.89) | 345.58 (150.13)

7. Secondary Outcome: ADAs
Description: Number of patients with antidrug antibodies after 3 months. Anti-erythropoietin antibodies screening was done using immunoprecipitation on the sample collected prior to the first dose of the first phase of the trial and on the 504-hour sample of the third phase
Time Frame: 120hr
Measure: Count of Participants; unit: Participants
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Anti-erythropoietin antibodies | 0 | 0 | 0
  No anti-erythropoietin antibodies detected | 24 | 24 | 24

8. Secondary Outcome: Adverse Events
Description: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Time Frame: 120hr
Measure: Count of Participants; unit: Participants
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Asthenia | 3 | 3 | 5
  Myalgia | 3 | 0 | 2
  Pruritus of trunk | 0 | 1 | 0
  Generalized myalgia | 0 | 1 | 1
  Arthralgia | 0 | 0 | 2
  Dorsal myalgia | 0 | 0 | 1
  Fracture | 1 | 0 | 1
  Headache | 2 | 0 | 0
  Pyrosis | 1 | 0 | 0
  Vomiting | 1 | 1 | 1
  Diarrhea | 0 | 0 | 1
  Nausea | 0 | 1 | 0
  No adverse events registered | 13 | 17 | 10

ADVERSE EVENTS:
Time Frame: The security profile was determined in all 3 periods of drug administration. All the volunteers were planned to received 3 doses of rhEPO. The duration of all clinical phase was 75 days. so, safety information was collected during 75 days.
Description: Adverse Event Reporting was conducted according to the regulation 6677/2010 (Section B.7) of the National Regulatory Agency
Arm/Group | Hemax® PFS 40,000 UI | Hemax® 40,000 UI | Erypo ® 40,000 UI
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 11/24 | 7/24 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemax® PFS 40,000 UI (N=24) | Hemax® 40,000 UI (N=24) | Erypo ® 40,000 UI (N=24)
Severe low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemax® PFS 40,000 UI (N=24) | Hemax® 40,000 UI (N=24) | Erypo ® 40,000 UI (N=24)
Asthenia (General disorders) | 3 (3) | 3 (3) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Pruritus of trunk (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dorsal myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is not allowed to disclose any confidential information of the clinical trial.